CLINICAL TRIAL: NCT04152226
Title: Clinical Study Protocol Number DBI-201- Open Label, Single-dose, Dose Escalating Evaluation of the Safety and Tolerability of DBI-001 in Patients With Tinea Pedis
Brief Title: A Trial to Evaluate the Safety and and Tolerability of DBI-001 in Patients With Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DBI-201
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Intervention Model Description: A single center open label dose escalating study design will be used in a population of patients with interdigital Tinea pedis. Each subject will have a single application of the test article applied to each foot. The three test articles will be a low dose, medium and a high dose of J. lividum. Each of the three groups will have 4 subjects. After the first cohort has completed their day 7 visits and if no significant tolerability of safety issues is identified the second cohort will be enrolled. After the second cohort has completed the day 7 visits and if no significant tolerability or safety issues are identified the third cohort will be enrolled. At all evaluations, signs and symptoms of application site reactions will be recorded at baseline, as well as days 2, 3, 7, 14, and 28.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Active Comparator): Cohort 1 DBI-001 Gel with 10^6 CFUs/ml of J.lividum
  Interventions: Drug: Janthinobacterium lividum
- Cohort 2 (Active Comparator): Cohort 2 DBI-001 Gel with 10^7 CFUs/ml of J.lividum
  Interventions: Drug: Janthinobacterium lividum
- Cohort 3 (Active Comparator): Cohort 3 DBI-001 Gel with 10^8 CFUs/ml of J.lividum
  Interventions: Drug: Janthinobacterium lividum

INTERVENTIONS:
Drug: Janthinobacterium lividum — Investigational Product

SUMMARY:
This is an open-label, single-dose, dose escalating evaluation of the safety and tolerability of three dose levels of DBI-001 in patients with Tinea pedis. The purpose of the current protocol is to establish the safety and tolerability of a single application of J. lividum to the feet of patients with proven T. pedis. In addition, the effect of J. lividum on the T. pedis will also be evaluated.

DETAILED DESCRIPTION:
Open-label, single-dose, dose escalating evaluation of the safety and tolerability of three dose levels of DBI-001 in patients with Tinea pedis. The test product will be applied by study personnel at the investigational site. Each subject will have a single application of approximately 0.5 ml of the test article applied to each foot. Both affected and unaffected feet will be treated covering the web spaces, toes, toe nails as well as the plantar and lateral aspect of both feet. Each of the three groups will have 4 subjects. After the first cohort has completed their day 7 visits, if no significant tolerability or safety issues identified the second cohort will be enrolled. After the second cohort has completed the day 7 visits and if no significant tolerability of safety issues is identified the third cohort will be enrolled.

ELIGIBILITY:
Subjects must meet all of the following criteria to be included in the study:

1. Witnessed, signed informed consent approved by Institutional Review Board/Independent Ethics Committee.
2. A signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of subject's individually identifiable health information.
3. Male Subjects of any race 18 years of age and older.
4. Subjects with a clinical diagnosis of interdigital T. pedis T. pedis interdigital defined as lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot (the non-interdigital lesions should not be hyperkeratotic, i.e., characteristic of tinea pedis moccasin).
5. Provisionally confirmed diagnosis at baseline by a positive potassium hydroxide (KOH) wet mount at the clinical site.
6. The sum of the clinical signs and symptoms scores of the target lesion is at least 4 using the Grading and signs and symptoms of T. pedis detailed in section 6.6.1, including a minimum score of at least 2 for erythema AND a minimum score of 2 for either scaling/fissures or pruritus/burning (on a scale of 0-3, where 2 indicates moderate severity). -

Exclusion Criteria:

Subjects with the following will be excluded from this study:

1. Any dermatological conditions that could interfere with clinical evaluations.
2. Any underlying disease(s) or some other dermatological condition that requires the use of interfering topical or systemic therapy.
3. Subjects that have not undergone the specified washout period(s) for the following topical preparations or subjects who require the concurrent use of any of the following topical medications applied to the foot: Topical astringents and abrasives (e.g. Burrow's solution) 1 week Topical antibiotics and antifungal on the infected area (e.g. Neomycin, Miconazole, Clotrimazole, Terbinafine) 2 weeks Anti-inflammatories, corticosteroids, topical immunomodulators (e.g. Pimecrolimus, Tacrolimus) 4 weeks
4. Subjects that have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications: Corticosteroids (including intramuscular injections) (e.g. Triamcinolone acetonide) 4 weeks Antibiotics (e.g. Tetracycline, Cephalosporins, etc.) and/or Antifungal agents (e.g. Fluconazole, Itraconazole, Terbinafine, etc.) 4 weeks Systemic immunomodulators (e.g. Cyclophosphamide, Azathioprine, Biologicals-Monoclonal Antibodies. 4 weeks
5. Treatment of any type of cancer within the last 6 months.
6. History of any significant internal disease (which contraindicates use of live microbiome e.g. leukemia, liver failure, cardiovascular disease)
7. Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
8. AIDS or AIDS related complex by medical history.
9. Known or suspected immune suppressive medications or diseases.
10. Diabetes mellitus Type I or II by medical history.
11. Peripheral vascular disease based on medical history.
12. Any subject not able to meet the study attendance requirements.
13. Subjects who have participated in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: : Daisy Blanco, MD, Study Director — Instituto Dermatologico y Cirugia de Piel
Locations (1):
- Instituto Dermatologico y Cirugia de Piel, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cohort 1 Dose 10^6CFUs/ml
  Janthinobacterium lividum: Investigational Product
- Cohort 2: Cohort 2 Dose 10^7CFUs/ml
  Janthinobacterium lividum: Investigational Product
- Cohort 3: Cohort 3 - Dose 10^8CFUs/ml
  Janthinobacterium lividum: Investigational Product
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Cohort 1 Dose 10^6CFUs/ml of J. lividum
  Janthinobacterium lividum: Investigational Product
- Cohort 2: Cohort 2 Dose 10^7CFUs/ml of J. lividum
  Janthinobacterium lividum: Investigational Product
- Cohort 3: Cohort 3 - Dose 10^8CFUs/ml of J. Lividum
  Janthinobacterium lividum: Investigational Product
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13.74) | 46.8 (3.3) | 35.8 (15.95) | 42.5 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 12
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 12
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation Cohort 1
Description: Tolerability will be evaluated through assessment of local signs and symptoms. For simplicity, as there were no local tolerability reactions, the cumulative tolerability, inclusive of Pruritus, Erythema, Edema, Scabbing/crusting, and Burning/Stinging is represented in the table. Scoring for of each Pruritus, Erythema, Edema, Scabbing/crusting, and Burning/Stinging according to the scoring system below. Tolerability events were only considered adverse events if they were grade 3 or higher or required discontinuation of test article or use of conmeds. As no Tolerability events satisfied this criteria, there were no tolerability associated adverse events.
  0 = none (complete absence)
  1. = mild (slight)
  2. = moderate (definitely present)
  3. = Severe
Time Frame: 28 days
Population: By number of feet treated
Measure: Count of Units; unit: Feet
Units Other Than Participants: Feet
Groups:
- 0=None Count n=24 (Percentage); 1=Mild Count n=24 (Percentage); 2=Moderate Count n=24 (Percentage); 3=Severe Count n=24: Symptom of Pruritus, Erythema, Edema, Scabbing/crusting, Burning/Stinging on areas unaffected by tinea pedis (by number of feet treated)
Arm/Group | 0=None Count n=24 (Percentage) | 1=Mild Count n=24 (Percentage) | 2=Moderate Count n=24 (Percentage) | 3=Severe Count n=24
Number analyzed (Participants) | 4 | 4 | 4 | 4
Number analyzed (Feet) | 8 | 8 | 8 | 8
Feet
  Pruritus Baseline | 8 | 0 | 0 | 0
  Pruritus 1 Hour Post application | 8 | 0 | 0 | 0
  Pruritus Day 2 | 8 | 0 | 0 | 0
  Pruritus Day 3 | 8 | 0 | 0 | 0
  Pruritus Day 7 | 8 | 0 | 0 | 0
  Pruritus Day 14 | 8 | 0 | 0 | 0
  Pruritus Day 28 | 8 | 0 | 0 | 0
  Erythema Baseline | 8 | 0 | 0 | 0
  Erythema 1 Hour Post | 8 | 0 | 0 | 0
  Erythema Day 2 | 8 | 0 | 0 | 0
  Erythema Day 3 | 8 | 0 | 0 | 0
  Erythema Day 7 | 8 | 0 | 0 | 0
  Erythema Day 14 | 8 | 0 | 0 | 0
  Erythema Day 28 | 8 | 0 | 0 | 0
  Edema Baseline | 8 | 0 | 0 | 0
  Edema 1 Hour Post | 8 | 0 | 0 | 0
  Edema Day 2 | 8 | 0 | 0 | 0
  Edema Day 3 | 8 | 0 | 0 | 0
  Edema Day 7 | 8 | 0 | 0 | 0
  Edema Day 14 | 8 | 0 | 0 | 0
  Edema Day 28 | 8 | 0 | 0 | 0
  Scabbing Baseline | 8 | 0 | 0 | 0
  Scabbing 1 Hour Post | 8 | 0 | 0 | 0
  Scabbing Day 2 | 8 | 0 | 0 | 0
  Scabbing Day 3 | 8 | 0 | 0 | 0
  Scabbing Day 7 | 8 | 0 | 0 | 0
  Scabbing Day 14 | 8 | 0 | 0 | 0
  Scabbing Day 28 | 8 | 0 | 0 | 0
  Pain Baseline | 8 | 0 | 0 | 0
  Pain 1 Hour Post | 8 | 0 | 0 | 0
  Pain Day 2 | 8 | 0 | 0 | 0
  Pain Day 3 | 8 | 0 | 0 | 0
  Pain Day 7 | 8 | 0 | 0 | 0
  Pain Day 14 | 8 | 0 | 0 | 0
  Pain Day 28 | 8 | 0 | 0 | 0

2. Primary Outcome: Safety Evaluation Cohort 2
Description: as for outcome 1
Time Frame: 28 days
Population: By number of feet treated
Measure: Count of Units; unit: Feet
Units Other Than Participants: Feet
Arm/Group | 0=None Count n=24 (Percentage) | 1=Mild Count n=24 (Percentage) | 2=Moderate Count n=24 (Percentage) | 3=Severe Count n=24
Number analyzed (Participants) | 4 | 4 | 4 | 4
Number analyzed (Feet) | 8 | 8 | 8 | 8
Feet
  Pruritus Baseline | 8 | 0 | 0 | 0
  Pruritus 1 Hour Post application | 8 | 0 | 0 | 0
  Pruritus Day 2 | 8 | 0 | 0 | 0
  Pruritus Day 3 | 8 | 0 | 0 | 0
  Pruritus Day 7 | 8 | 0 | 0 | 0
  Pruritus Day 14 | 8 | 0 | 0 | 0
  Pruritus Day 28 | 8 | 0 | 0 | 0
  Erythema Baseline | 8 | 0 | 0 | 0
  Erythema 1 Hour Post | 8 | 0 | 0 | 0
  Erythema Day 2 | 8 | 0 | 0 | 0
  Erythema Day 3 | 8 | 0 | 0 | 0
  Erythema Day 7 | 8 | 0 | 0 | 0
  Erythema Day 14 | 8 | 0 | 0 | 0
  Erythema Day 28 | 8 | 0 | 0 | 0
  Edema Baseline | 8 | 0 | 0 | 0
  Edema 1 Hour Post | 8 | 0 | 0 | 0
  Edema Day 2 | 8 | 0 | 0 | 0
  Edema Day 3 | 8 | 0 | 0 | 0
  Edema Day 7 | 8 | 0 | 0 | 0
  Edema Day 14 | 8 | 0 | 0 | 0
  Edema Day 28 | 8 | 0 | 0 | 0
  Scabbing Baseline | 8 | 0 | 0 | 0
  Scabbing 1 Hour Post | 8 | 0 | 0 | 0
  Scabbing Day 2 | 8 | 0 | 0 | 0
  Scabbing Day 3 | 8 | 0 | 0 | 0
  Scabbing Day 7 | 8 | 0 | 0 | 0
  Scabbing Day 14 | 8 | 0 | 0 | 0
  Scabbing Day 28 | 8 | 0 | 0 | 0
  Pain Baseline | 8 | 0 | 0 | 0
  Pain 1 Hour Post | 8 | 0 | 0 | 0
  Pain Day 2 | 8 | 0 | 0 | 0
  Pain Day 3 | 8 | 0 | 0 | 0
  Pain Day 7 | 8 | 0 | 0 | 0
  Pain Day 14 | 8 | 0 | 0 | 0
  Pain Day 28 | 8 | 0 | 0 | 0

3. Primary Outcome: Safety Evaluation Cohort 3
Description: as for outcome 1
Time Frame: 28 days
Population: By number of feet treated
Measure: Count of Units; unit: Feet
Units Other Than Participants: Feet
Arm/Group | 0=None Count n=24 (Percentage) | 1=Mild Count n=24 (Percentage) | 2=Moderate Count n=24 (Percentage) | 3=Severe Count n=24
Number analyzed (Participants) | 4 | 4 | 4 | 4
Number analyzed (Feet) | 8 | 8 | 8 | 8
Feet
  Pruritus Baseline | 8 | 0 | 0 | 0
  Pruritus 1 Hour Post application | 8 | 0 | 0 | 0
  Pruritus Day 2 | 8 | 0 | 0 | 0
  Pruritus Day 3 | 8 | 0 | 0 | 0
  Pruritus Day 7 | 8 | 0 | 0 | 0
  Pruritus Day 14 | 8 | 0 | 0 | 0
  Pruritus Day 28 | 8 | 0 | 0 | 0
  Erythema Baseline | 8 | 0 | 0 | 0
  Erythema 1 Hour Post | 8 | 0 | 0 | 0
  Erythema Day 2 | 8 | 0 | 0 | 0
  Erythema Day 3 | 8 | 0 | 0 | 0
  Erythema Day 7 | 8 | 0 | 0 | 0
  Erythema Day 14 | 8 | 0 | 0 | 0
  Erythema Day 28 | 8 | 0 | 0 | 0
  Edema Baseline | 8 | 0 | 0 | 0
  Edema 1 Hour Post | 8 | 0 | 0 | 0
  Edema Day 2 | 8 | 00 | 0 | 0
  Edema Day 3 | 8 | 0 | 0 | 0
  Edema Day 7 | 8 | 0 | 0 | 0
  Edema Day 14 | 8 | 0 | 0 | 0
  Edema Day 28 | 8 | 0 | 0 | 0
  Scabbing Baseline | 8 | 0 | 0 | 0
  Scabbing 1 Hour Post | 8 | 0 | 0 | 0
  Scabbing Day 2 | 8 | 0 | 0 | 0
  Scabbing Day 3 | 8 | 0 | 0 | 0
  Scabbing Day 7 | 8 | 0 | 0 | 0
  Scabbing Day 14 | 8 | 0 | 0 | 0
  Scabbing Day 28 | 8 | 0 | 0 | 0
  Pain Baseline | 8 | 0 | 0 | 0
  Pain 1 Hour Post | 8 | 0 | 0 | 0
  Pain Day 2 | 8 | 0 | 0 | 0
  Pain Day 3 | 8 | 0 | 0 | 0
  Pain Day 7 | 8 | 0 | 0 | 0
  Pain Day 14 | 8 | 0 | 0 | 0
  Pain Day 28 | 8 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Description: Treatment-emergent adverse events are those with onset after application. Related defined as "Definitely", "Probably", or "Possibly". Not Related defined as "Unlikely" or "None".
  Tolerability events were only considered adverse events if they were grade 3 or higher or required discontinuation of test article or use of conmeds. As no Tolerability events satisfied this criteria, there were no tolerability associated adverse events.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04152226/Prot_SAP_000.pdf